CLINICAL TRIAL: NCT03492957
Title: PHysical Activity for Non-ambulatory Stroke Survivors (PHANSS-2): Developing a Feasible and Acceptable Intervention for Stroke Survivors Who Cannot Walk Independently
Brief Title: PHysical Activity for Non-ambulatory Stroke Survivors: Feasibility Study
Acronym: PHANSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Edinburgh (Other); Edinburgh Napier University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHLS1
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: physical activity; exercise; non-ambulatory; feasibility; mixed methods
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants can select either individual treatment at home, or group treatment in a community setting, but the intervention content and dose are the same.
Masking Description: Blinding: outcomes are assessed by independent assessors, otherwise not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): A tailored, person-centred, 12-week, chair-based exercise intervention to increase physical activity and fitness. Dose: one face-face session with a qualified physiotherapist plus two independent sessions per week. This is combined with education on self-management, self-efficacy and lifestyle change. There is no control group ion this feasibility study.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — A tailored, person-centred, 12-week, chair-based exercise intervention to increase physical activity and fitness. Dose: one face-face session with a qualified physiotherapist plus two independent sessions per week. This is combined with education on self-management, self-efficacy and lifestyle change.
  Other Names: Education on self-management, self-efficacy and lifestyle

SUMMARY:
The aim of this study is to design a physical activity programme for non-ambulatory stroke survivors (delivered via either community-based groups or a home-based individual programme) and evaluate its feasibility, acceptability, preliminary and adverse effects. The study will also explore the views of non-ambulatory stroke survivors and their carers on: needs, personal goals, barriers, and motivators, experiences of programme participated in and preferred format (i.e. home-based individual/ community-based groups).

DETAILED DESCRIPTION:
Background:

Physical activity interventions after stroke are needed because stroke survivors are under-active; their average physical fitness level is about 50% of sedentary healthy controls. This adversely affects vascular risk factor profiles, disability and participation, problems that are all likely to be exacerbated in stroke survivors who are unable to walk. Fitness can be improved after stroke through cardiorespiratory training. This also improves psychosocial functioning and adaptation to life after stroke. Community-based services for exercise after stroke are developing throughout the UK. However, current evidence, associated guidelines and exercise professional training mainly pertain to ambulatory stroke survivors; non-ambulatory stroke survivors have hardly been involved in this area of research. In this study, we define "non-ambulatory" as requiring at least "continuous or intermittent support of one person to help with balance or coordination" (i.e. Functional Ambulatory Category ≤ 2).

Study aim:

The aim of this study is to design a physical activity programme for non-ambulatory stroke survivors (delivered via either community-based groups or a home-based individual programme) and evaluate its feasibility, acceptability, preliminary and adverse effects. The study will also explore the views of non-ambulatory stroke survivors and their carers on: needs, personal goals, barriers, and motivators, experiences of programme participated in and preferred format (i.e. home-based individual/ community-based groups).

Study design:

Mixed-methods, observational feasibility study. This study will incorporate qualitative interviews/focus groups to explore the experiences of the programme participants are taking part in and their thoughts and views of PA after stroke. Interviews and focus groups will be conducted throughout the physical activity programme.

Participant recruitment:

Participants will be recruited by the Scottish Stroke Research Network (SRN) via: databases and electronic patient medical/nursing/AHP notes, records of discharges from acute stroke wards to off-site rehabilitation units and word of mouth among AHPs., within NHS Lanarkshire.

Participants will also be recruited via non-NHS sites: local community stroke groups, social media, stroke charities, press releases and related media and care homes.

Study setting:

Glasgow Caledonian University will be used for the community-based group programme and focus groups/interviews.

Participants' own home setting will be used for the home-based, individual programme and interviews.

Study participants:

Non-ambulatory stroke survivors and their carers (where applicable) living at home or in care homes.

Study outcomes:

Outcomes will include measures of disability, ADL, strength, anxiety and depression, sedentary behaviour, self-efficacy, health status, attainment of individual goals, as well as carer burden (where appropriate).

Feasibility will be assessed by numbers of participants invited to participate, accepting and being recruited into the study, completing the intervention, programme adherence and drop outs. Safety data will be examined using data on adverse effects reported by participants.

Study duration: 12 months.

ELIGIBILITY:
Inclusion Criteria (stroke survivors):

* Age 18 years or over
* Clinical diagnosis of stroke
* Non-ambulatory, defined as requiring at least "continuous or intermittent support of one person to help with balance or coordination" (i.e. Functional Ambulatory Category ≤ 2) most of the time.
* Able to give informed consent (by proxy if appropriate)
* Able to travel via private taxi to community venue (for group exercise, if preferred)
* For care home residents: participant must not be participating in any structured form of PA run within their care home.
* Participant residing in private home or care home (must be discharged from in-patient care at start of intervention)

Exclusion Criteria (stroke survivors):

* Judged by treating GP to be too unwell to participate
* Uncontrolled medical condition that contraindicates exercise e.g. uncontrolled cardiac condition
* Severe cognitive impairment (unable to follow and understand instructions)

Inclusion criteria (carers):

- Able to give informed consent

Exclusion criteria (carers):

- Not well enough to participate (as per self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 3-month follow-up
  Person-centred tool for goal setting and evaluation

SECONDARY OUTCOMES:
Barthel Index (BI) | 3-month follow-up
  Measure to evaluate independence in activities of daily living
Stroke Impact Scale (SIS) | 3-month follow-up
  Measure to evaluate impact of intervention on stroke-related impairments, activity limitations and participation restrictions
Stroke Self-Efficacy questionnaire (SSEQ) | 3-month follow-up
  Measure to evaluate level of confidence
Hospital Anxiety and Depression Scale (HADS) | 3-month follow-up
  Measure to evaluate levels of anxiety and depression
Motricity Index (MI) | 3-month follow-up
  Clinical evaluation of muscle strength in both affected and non-affected upper and lower limbs
Force measurements | 3-month follow-up
  Quantitative measurements of muscle force in quadriceps and hamstring muscles in both affected and unaffected lower limbs using dynamometry
Caregiver Burden Scale (CBS) | 3-month follow-up
  A questionnaire to evaluate carer burden
Activity data | 3-month follow-up
  Quantitative data from an activity monitor to measure sedentary behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Frederike MJ van Wijck, PhD, Principal Investigator — Glasgow Caledonian University

IPD SHARING:
Plan to Share IPD: Undecided